CLINICAL TRIAL: NCT05661851
Title: Clinical Evaluation of a Multidose Preservative-free Lubricating Eye Drops Contained in Novelia® Eye Dropper in Non-Contact Lens Wearing Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR-6502
Record Dates: First submitted 2022-12-14; First posted 2022-12-22 (Actual); Results first posted 2024-05-01 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Investigational product (Experimental): Eligible subjects will be randomly assigned the investigational product to be used in both eyes for the duration of the study.
  Interventions: Drug: Investigational Lubricating Eye Drop in a Novelia® bottle
- Control product (Active Comparator): Eligible subjects will be randomly assigned the control product to be used in both eyes for the duration of the study
  Interventions: Drug: Blink® Tears eye Drops

INTERVENTIONS:
Drug: Investigational Lubricating Eye Drop in a Novelia® bottle — Investigational Product
  Arms: Investigational product
Drug: Blink® Tears eye Drops — Control Product
  Arms: Control product

SUMMARY:
This is a 30-Day, multi-site, single-masked, bilateral, active- controlled, 2-Arm parallel group study to evaluate the safety and efficacy of an Investigational product.

ELIGIBILITY:
Inclusion Criteria:

Potential subjects must satisfy all of the following criteria to be enrolled in the study:

1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. Be between 18 and 69 (inclusive) years of age at the time of screening.
4. Possess a wearable pair of spectacles that provide correction for distance vision and bring them to every visit (only if applicable- to the investigator's discretion).
5. Self-reported symptoms of ocular dryness and/or the use of artificial tears in the last 3 months.
6. Subjects must be non-contact lens wearers.
7. The best corrected, monocular, distance visual acuity must be 20/30 or better in each eye, either unaided or best corrected.

Exclusion Criteria:

Potential subjects must satisfy all of the following criteria to be enrolled in the study:

1. Be currently pregnant or lactating.
2. Be diabetic.
3. Be currently using any ocular medications or have any ocular infection of any type which may interfere with the clinical trial (at the investigator's discretion).
4. By self-report, have any ocular or systemic disease, allergies, infection, or use of medication that might contraindicate or interfere with the clinical trial, or otherwise compromise study endpoints, including infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive disease (e.g., Human Immunodeficiency Virus [HIV]), autoimmune disease (e.g., rheumatoid arthritis, Sjögren's syndrome), or history of serious mental illness or seizures. See section 9.1 for additional details regarding excluded systemic medications.
5. Have habitually worn rigid gas permeable (RGP) lenses, orthokeratology lenses, or hybrid lenses (e.g., SynergEyes, SoftPerm) within the past 3 months and soft contact lenses in the past 1 month.
6. Have participated in any pharmaceutical or medical device related clinical trial within 30 days prior to study enrollment.
7. Be an employee (e.g., Investigator, Coordinator, Technician) or immediate family member of an employee (including partner, child, parent, grandparent, grandchild or sibling of the employee or their spouse) of the clinical site.
8. Be a current habitual user of prescription medication to treat dry eye and ocular discomfort, ocular steroids, or any medication (RX or OTC), except for artificial tears that would interfere with the clinical study (at the discretion of the investigator).
9. Have any known allergy or sensitivity to ingredients that the investigational product may contain (e.g., Sodium Chlorite, Boric Acid, Sodium Borate Decahydrate, Sodium Chloride, Potassium Chloride, Calcium Chloride Dihydrate, Magnesium Chloride Hexahydrate, Polyethylene Glycol 400, Sodium Hyaluronate and Purified Water).
10. Have clinically significant (grade 3 or higher on the FDA grading scale) slit lamp findings (e.g., corneal edema, neovascularization or staining, tarsal abnormalities, or bulbar injection) or other corneal or ocular disease or abnormalities that contraindicate participation or may otherwise compromise study endpoints (including entropion, ectropion, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, moderate or above corneal distortion, herpetic keratitis).
11. Have a history of strabismus or amblyopia.
12. Have had or have planned (within the study period) any ocular or intraocular surgery (e.g., radial keratotomy, PRK, LASIK, iridotomy, cataract removal, retinal laser photocoagulation, etc.).
13. Have any significant corneal distortion due to previous contact lens wear, surgery, or pathology (At the discretion of the investigator).

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2023-02-23 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (8):
- United States (8):
  - Vue Optical Boutique, Jacksonville, Florida
  - Stam & Associates Eye Care, Jacksonville, Florida
  - Kannarr Eye Care, Pittsburg, Kansas
  - Complete Eye Care of Medina, Medina, Minnesota
  - ProCare Vision Centers, Granville, Ohio
  - Total Eye Care, Memphis, Tennessee
  - Tyler Eye Associates, Tyler, Texas
  - Botetourt Eyecare, LLC, Salem, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 121 subjects were enrolled in this study. Of those enrolled, 118 subjects were dispensed at least one study eyedrop while 3 subjects failed to meet all eligibility criteria. Of those dispensed, 107 subjects completed the study while 11 subjects were discontinued.
Groups:
- Test: Subjects that were randomized to the Test group throughout the duration of the study.
- Control: Subjects that were randomized to the Control group throughout the duration of the study.
Period: Overall Study
Arm/Group | Test | Control
Started | 58 | 60
Completed | 53 | 54
Not Completed | 5 | 6
Not completed — Protocol Violation | 1 | 1
Not completed — Covid-19 Related | 3 | 4
Not completed — investigational product Was Dispensed Incorrectly At Visit 2 | 1 | 0
Not completed — The Patient Was Dispensed The Incorrect investigational product At Visit 2 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All subjects dispensed at least one study eyedrop.
Groups:
- Total: Total of all reporting groups
Arm/Group | Test | Control | Total
Number analyzed (Participants) | 58 | 60 | 118
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.2 (14.23) | 50.1 (13.79) | 49.2 (13.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 41 | 86
  Male | 13 | 19 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 3 | 2 | 5
  Black or African American | 8 | 6 | 14
  White | 45 | 51 | 96
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Overall Quality of Ocular Comfort From Baseline to 30-Day Follow-Up Using VAS Scores
Description: Subjective ocular comfort was assessed at baseline, and at 30-day follow-up using a Visual Analogue Scale (VAS) with continuous scale from 0 (extremely uncomfortable) to 100 (extremely comfortable). The change from baseline ocular comfort score was calculated as 30-day follow-up score minus baseline score. Change from baseline VAS scores range from -100 to 100, where higher change from baseline comfort scores indicates better performance. The average change from baseline comfort score for each Arm was reported.
Time Frame: Baseline and 30-Day Follow-up
Population: All randomized subjects regardless of actual treatment and subsequent withdrawal from the study or deviation from the protocol.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Test | Control
Number analyzed (Participants) | 53 | 54
Scores on a scale | 18.47 (22.125) | 9.65 (22.859)
Statistical Analysis 1: Comparison: Test vs Control; A sample size of 104 subjects provides at least 90% statistical power to test non-inferiority of the Test eyedrop compared to the Control eyedrop using a two sample t-test with a two-sided type I error rate of 0.05; Test type: Non-Inferiority — Non-inferiority margin of -20 was used; Linear Mixed Model; Kenward and Roger Method was used for the denominator degrees of freedom; Least-square Mean Difference = 5.9, 95% CI 2-sided [-1.67 to 13.38], Standard Error of Mean 3.79 — LS Mean difference was calculated as Test minus Control

2. Secondary Outcome: Change in Overall Quality of Vision From Baseline to 30-Day Follow-Up Using VAS Scores
Description: Subjective vision was assessed at baseline, and at 30-day follow-up using a Visual Analogue Scale (VAS) with continuous scale from 0 (extremely uncomfortable) to 100 (extremely comfortable). The change from baseline quality of vision score was calculated as 30-day follow-up score minus baseline score. Change from baseline VAS scores range from -100 to 100, where higher change from baseline vision scores indicates better performance. The average change from baseline vision score for each arm was report.
Time Frame: Baseline and 30-Day Follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Test | Control
Number analyzed (Participants) | 53 | 54
Scores on a scale | 11.55 (22.863) | 5.70 (23.615)
Statistical Analysis 1: Comparison: Test vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — Non-inferiority margin of -20 was used; Bootstrapping methods; Mean Population Difference Estimate = 5.843, 95% CI 2-sided [-2.8904 to 14.5768], Standard Error of Mean 4.4560 — Bootstrap Mean Difference was calculated as Test minus Control

ADVERSE EVENTS:
Time Frame: Throughout the entire duration of the study. Approximately 30 Days per subject.
Arm/Group | Test | Control
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/60
Other Adverse Events (participants affected / at risk) | 0/58 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-25): https://cdn.clinicaltrials.gov/large-docs/51/NCT05661851/Prot_SAP_000.pdf